CLINICAL TRIAL: NCT06169449
Title: Weight Management in Overweight Endometrial Cancer Patients Undergoing Fertility-sparing Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaodan Li, Director, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDL2022-49
Record Dates: First submitted 2023-11-12; First posted 2023-12-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Endometrium Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weight management Group (Experimental): Patients in the weight management group used a weight management model that included diet, exercise, accompany and refresh.
  Interventions: Behavioral: Weight management--diet; Behavioral: Weight management--exercise; Behavioral: Weight management--accompany; Behavioral: Weight management--refresh
- Control Group (Other): Patients in the control group underwent routine care for self-weight management.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Weight management--diet — The diet structure adopts an energy-limited balanced diet. In this structure, the total daily energy intake is reduced by 500~1000 kcal based on the target energy intake; however, the balance is maintained for the energy supply ratio of the three major nutrients (with carbohydrate, protein, and fat accounting for 55~60%, 10~20%, and 15~30% of the total daily energy, respectively). Combined with the patient's eating habits, the food exchange portion method is used as a guide; each portion providing 90 kcal is considered as one portion. Specific recipes are formulated after calculating the ideal weight and the total daily calorie intake based on activity intensity, determining the number of six food exchange portions and the distribution of three meals according to the total calorie and diet structure, and combining the equivalent food exchange table based on individual tastes and preferences; this ensures patient acceptability and implementation.
  Arms: Weight management Group
Behavioral: Weight management--exercise — Exercise goals are divided into four levels based on individual health conditions and personal preferences; these include: cultivating exercise habits, improving cardiopulmonary function, enhancing muscle strength, and improving flexibility. Individualized exercise prescriptions that specify the exercise type, intensity, time, and frequency are formulated.
  Arms: Weight management Group
Behavioral: Weight management--accompany — This component involves the inclusion of patients in online management. Online groups are established, daily feedback is obtained regarding weight management implementation, self-sharing is encouraged, and peer support is established; a total of 6 sessions of online health education are provided once every 4 weeks for 20-60 minutes at each session. This includes information regarding the risks associated with overweightness and obesity; weight management benefits; knowledge regarding diet and nutrition, exercise and sports, and behavioral styles; and problem exchange and sharing, among others. Professional support is provided by weekly communication with patients one-on one via WeChat or telephonic conversations. The patient's diet and exercise record sheet are checked, patients are asked questions regarding implementation of the current program and any discomfort or difficulties; corresponding guidance is provided as appropriate.
  Arms: Weight management Group
Behavioral: Weight management--refresh — According to the dietary nutrition guidelines for Chinese residents, patients are advised to drink 2500 ml or more of water daily; they are also advised to work and rest regularly to ensure sufficient sleep time, ensure smooth bowel movements, take deep breaths when waking up in the morning, pay attention to the work-rest balance, avoid being sedentary, and stand up and move around at least once every 50 minutes, maintain physical vitality by adjusting daily living habits.
  Arms: Weight management Group
Behavioral: Control group — The relationship between overweightness and obesity and endometrial cancer risk was explained to patients in the control group and their willingness for self-weight management was respected. Communication was maintained with patients from treatment initiation to 3 and 6 months after treatment; patients' questions regarding weight reduction were answered and suggestions were provided regarding nutrition, exercise, and lifestyle management.
  Arms: Control Group

SUMMARY:
In this study, overweight and obese patients with endometrial cancer treated with fertility- sparing therapy were randomly divided into two groups. The test group was given weight management, while the control group was given routine care. Relevant information such as body morphology and composition, glycolipid metabolism, molecular typing and tumor outcomes of the subjects were collected. By evaluating the tumor outcome and changes in glycolipid metabolism indicators, to confirm the effectiveness and safety of weight management for overweight and obese patients with endometrial cancer and treatd with fertility preservation.

DETAILED DESCRIPTION:
Obesity is recognized as a major risk factor for the development of endometrial cancer. Notably, several retrospective studies have shown that obesity reduces complete remission and pregnancy rates and increases recurrence rates in patients with endometrial cancer and atypical hyperplasia who undergo fertility-sparing treatment. Guidelines or consensus statements for fertility-sparing treatment in endometrial cancer recommend weight management. However, prospective intervention studies on the effectiveness of systematic weight management models in patients receiving reproductive function-preserving treatment for endometrial cancer and atypical hyperplasia are lacking. This study therefore aimed to investigate the impact of the weight management on body morphology and composition, glycolipid metabolism, and tumor outcomes in overweight and obese patients with endometrial cancer and atypical hyperplasia who underwent reproductive function-preserving treatments.In this study, overweight and obese patients with endometrial cancer treated with fertility- sparing therapy were randomly divided into two groups. The test group was given weight management, while the control group was given routine care. Relevant information such as body morphology and composition, glycolipid metabolism, molecular typing and tumor outcomes of the subjects were collected. By evaluating the tumor outcome and changes in glycolipid metabolism indicators, to confirm the effectiveness and safety of weight management for overweight and obese patients with endometrial cancer and treatd with fertility preservation.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years old
* diagnosed as endometrial cancer or atypical hyperplasia
* immunohistochemical staining and sequencing of pathological tissue
* fertility-preserving therapy
* BMI≥25 kg/m2
* informed consent.

Exclusion Criteria:

* those with communication barriers
* pregnant women
* medical and surgical serious complications: urinary calculi, history of renal failure or severe renal insufficiency, familial dyslipidemia, severe liver disease, chronic metabolic acidosis, history of pancreatitis, severe diabetes mellitus, active gallbladder disease, fat dyspepsia, severe cardiovascular and cerebrovascular diseases.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index（BMI）--physiological parameter | 6 months of intervention
  Use the Inbody720 to measure height and weight and calculate BMI according to the formula"BMI (= weight (kg)/height2 (m2)"
waist-to-height ratio (WHtR)--physiological parameter | 6 months of intervention
  Calculate WHtR according to the formula"WHtR= waist circumference (cm)/height (cm)= waist circumference (cm)/height (cm)"
waist-to-hip ratio (WHR)--physiological parameter | 6 months of intervention
  Calculate WHR according to the formula"WHR=waist circumference (cm)/hip circumference (cm)"
body shape index (ABSI)--physiological parameter | 6 months of intervention
  Calculate ABSI according to the formula"ABSI= (waist)/([BMI]^2/3×height^1/2)"
body roundness index (BRI)--physiological parameter | 6 months of intervention
  Calculate BRI according to the formula"BRI= waist/BMI"
visceral fat index (VAI)--physiological parameter | 6 months of intervention
  Calculate VAI according to the formula"VAI= waist/(36.58 + 1.89 × BMI) × triglyceride (TG) level/0.81 × 1.52/high density lipoprotein (HDL) level"
lipid accumulation index (LAP) (female)--physiological parameter | 6 months of intervention
  Calculate LAP according to the formula"LAP= = (waist circumference - 58) × TG level"
waist circumference--physiological parameter | 6 months of intervention
  measured with the subject's body upright, abdomen relaxed, both arms hanging down naturally, feet together, and the tape measure placed around the waist; the height was adjusted to the horizontal plane passing through the midpoint of the line between the lower edge of the rib arch and the iliac crest in the mid-axillary line
hip circumference--physiological parameter | 6 months of intervention
  measured with the subject's body upright, taking the circumference of the body at the horizontal position of the uppermost point of the hip
body fat mass (BFM)--physiological parameter | 6 months of intervention
  Measured by the Inbody720 Human Body Composition Analyzer
muscle mass--physiological parameter | 6 months of intervention
  Measured by the Inbody720 Human Body Composition Analyzer
percent body fat (PBF)--physiological parameter | 6 months of intervention
  Measured by the Inbody720 Human Body Composition Analyzer
basal metabolic rate--physiological parameter | 6 months of intervention
  Measured by the Inbody720 Human Body Composition Analyzer
visceral fat area (VFA)--physiological parameter | 6 months of intervention
  Measured by the Inbody720 Human Body Composition Analyzer
triglycerides--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
cholesterol--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
high density lipoprotein(HDL)--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
low density lipoprotein--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
fasting glucose--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
fasting insulin (FINS)--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
glycated hemoglobin--physiological parameter | 6 months of intervention
  About 5 ml of venous blood was drawn from the study subjects in the fasting state in the morning and sent to the Laboratory Department of the People's Hospital of Peking University, where it was measured by Beckman AU5800 biochemical analyzer.
homeostatic model assessment of insulin resistance (HOMA-IR) index--physiological parameter | 6 months of intervention
  Calculate HOMA-IR according to the formula"HOMA-IR= fasting blood glucose (mmol/L) × FINS level (mU/mL)/22.5"

SECONDARY OUTCOMES:
Complete remission | 6 months of intervention
  Complete remission indicated by complete endometrial regression and interstitial metaplasia-like changes on histopathology after treatment (without any endometrial atypical hyperplasia or endometrioid adenocarcinoma lesions, as clarified by pathologists)
Recurrence | 6 months of intervention
  After complete remission, the reappearance of endometrioid adenocarcinoma or atypical endometrial hyperplasia during follow-up or after pregnancy or childbearing is defined as recurrence and is diagnosed by the pathologist.
Pregnancy | 2 years of intervention
  The clinical diagnosis was pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaodan Li, Master, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China, China

REFERENCES:
- [Derived] Chen Y, Yang J, Wan Y, Li Q, Yang D, Wang Y, Gong J, Bai L, Liu Y, Li X, Wang J. DEAR model in overweight endometrial cancer patients undergoing fertility-sparing treatment: A randomized controlled trial. Gynecol Oncol. 2024 Jun;185:148-155. doi: 10.1016/j.ygyno.2024.02.017. Epub 2024 Feb 28. PMID 38422947